CLINICAL TRIAL: NCT00414414
Title: A Randomized, Prospective Double Blind Placebo Control Clinical Trial of Prednisone as Adjunctive Therapy for the Treatment of Hospitalized Patients With Pulmonary TB and HIV Co-infection
Brief Title: A RCT of Prednisone as Adjunctive Therapy for Hospitalized Patients With Pulmonary TB and HIV Co-infection
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding not awarded
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006301-01H
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2010-08

CONDITIONS: Tuberculosis; HIV Infections
Keywords: TB; Tuberculosis; HIV; Co-infection; Steroid; Prednisone; oral corticosteroids; TB Treatment; South Africa
MeSH Terms: conditions — Tuberculosis; HIV Infections; Coinfection | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- prednisone (Active Comparator)
  Interventions: Drug: Prednisone
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Prednisone
  Other Names: non applicable
  Arms: prednisone
Drug: placebo — placebo
  Other Names: non applicable
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if 30-day survival will be improved with addition of prednisone to standard tuberculosis (TB) therapy.

DETAILED DESCRIPTION:
Tuberculosis (TB) is the leading cause of death in people infected with HIV worldwide. South Africa has one of the highest rates of tuberculosis and HIV in sub Saharan Africa and the world. Infection with HIV can result in activation of the latent form of TB to its active form. In places like sub Saharan Africa where the HIV rates are very high TB has spread with incredible vigor. In order to study this phenomenon, we conducted a preliminary project, which demonstrated that there are approximately 250 patients with active TB admitted to one urban South African hospital in one month and that almost half of them are infected with HIV. One quarter of them died while in hospital. They were young people with an average of 32 years. We are interested in undertaking clinical trials that will study novel therapies that can be added to the existing antimicrobial regimens in order to reduce the number of people dying from TB. One of these therapies would be the addition of prednisone, an oral steroid, to the standard TB treatment regimen. Steroids have been shown to be useful in TB meningitis and pericarditis in HIV positive and negative patients. However, steroids have never been tested in a formal manner in HIV patients with pulmonary TB. We have chosen to do our research in South Africa since the numbers of patients needed to design a clinical trial such as the one presented can only be found in such an environment. Prednisone is cheap, easily obtainable and thus a sustainable intervention in developing countries. The impact of the research would affect not only the international community including Canada but would certainly have a lasting sustainable effect on the local community in Pietermaritzburg, South Africa in addition to the rest of the world.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AFB smear positive pulmonary TB (via microscopy)
* must be on quadruple standard chemotherapy for TB
* patients admitted to the medical ward (Edendale Hospital (EDH)- Pietermaritzburg,KwaZulu Natal, South Africa)
* must survive the first 24 hours after admission. In addition it takes up to 24 hours for the lab to assess all of the sputum samples sent for analysis
* patients must live in Pietermaritzburg in order to ensure efficient follow up
* positive HIV test (new or documented serodiagnosis via HIV antibody testing (ELISA Bio-rad ACCESS HIV 1/2 Immunoassay System))*
* adults >17 yrs of age
* consent to enter study * Only a screening test will be done to identify HIV positive patients, as the high prevalence of HIV in patients with pulmonary TB (60%) results in a very high positive predictive value, and a Western blot would not be needed as a confirmatory test.

Exclusion Criteria:

* TB meningitis *
* TB pericarditis *
* adrenal Insufficiency *
* old tuberculosis (Treatment for > 1 month prior to admission, Treatment failure) or known MDR-TB
* significant co-morbidities such as diabetes, uncontrolled HTN, peptic ulcer disease and renal disease and palliative conditions (untreatable cancer), or another infection
* other serious HIV related diseases such as cryptococcal meningitis, and Non Hodgkin's Lymphoma
* pregnancy
* previously treated with corticosteroids in the last month prior to admission, (9) other pulmonary pathogens identified in sputum 10) allergy to co-trimoxazole) (refer to co-trimoxazole section) *Based on clinical evaluation these patients will be excluded because evidence exists for using steroids in these conditions.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Our primary objective is to determine if 30-day survival will be improved with addition of prednisone to quadruple standard TB therapy. We will measure all cause mortality at 30 days. | 30 days

SECONDARY OUTCOMES:
Our secondary endpoints will involve the measurement of clinical, laboratory and radiological parameters and adverse reactions. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Alvarez, MD, Study Chair — Ottawa Hospital Research Institute
Locations (2):
- The Ottawa Hospital - General Campus, Ottawa, Ontario, Canada
- Erendale Hospital, Pietermaritzburg, KwaZulu-Natal, South Africa